CLINICAL TRIAL: NCT05321901
Title: Effects of a Telerehabilitation Program Based on Biopsychosocial Approach in Women With Rheumatic Disease
Brief Title: Telerehabilitation in Women With Rheumatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Erkin Oğuz SARI, Principal Investigator, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/106
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Rheumatic Disease
Keywords: Rheumatic diseases; Telerehabilitation; Chronic pain; COVID-19; Biopsychosocial Approach
MeSH Terms: conditions — Rheumatic Diseases; Chronic Pain; COVID-19 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Telerehabilitation assisted exercise program (Active Comparator): The telerehabilitation-assisted exercise program included a Biopsychosocial Exercise Therapy approach (BETY).
  The approaches that make up the BETY innovation are grouped under 4 headings: Patient education on chronic pain, functional body stabilization exercises (mind-body information management), dance therapy-authentic movement (emotion-state information management), and sexual information management.
  Tele-rehabilitation group participated in the sessions that lasted for one and a half hours, 3 days a week for 8 weeks, over the Whatsapp group.
  The investigators, who provided supervision during the sessions, also participated in the exercises simultaneously.
  Interventions: Other: Biopsychosocial Exercise Therapy approach (BETY)
- Control Group (Other): The control group participants were those who did not want to receive exercise treatment with telerehabilitation and took their routine medications during the 8 weeks period.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Biopsychosocial Exercise Therapy approach (BETY) — The BETY intervention is grouped under 4 headings: Patient education on chronic pain, functional body stabilization exercises (mind-body information management), dance therapy-authentic movement (emotion-state information management), and sexual information management.
  Arms: Experimental Group: Telerehabilitation assisted exercise program
Other: Control group — The control group participants were those who did not want to receive exercise treatment with telerehabilitation and took their routine medications during the 8 weeks period.
  Arms: Control Group

SUMMARY:
This study aims to investigate the effectiveness of the Biopsychosocial Exercise Therapy Approach (BETY), which is a biopsychosocial model, on daily living activities, anxiety, depression, and biopsychosocial conditions through telerehabilitation in rheumatic patients who could not go to the clinics during the COVID-19 pandemic.

DETAILED DESCRIPTION:
35 female participants with rheumatic disease were included in the study. Among the individuals who participated in face-to-face BETY sessions before, 23 individuals who agreed to exercise with telerehabilitation were divided into 2 groups, the exercise group, and 12 individuals in the control group.

Group 1: Telerehabilitation group: Individuals in the telerehabilitation group attended sessions that lasted for one and a half hours, 3 days a week for 8 weeks, in the company of a physiotherapist over the Whatsapp group. The investigators, who provided supervision during the sessions, also participated in the exercises simultaneously. The investigators managed the individuals according to their exercise number and order, by reminding them of the exercises with explanatory messages and positive energy via Whatsapp group. The participation of the patients in the exercises was followed up with the answers they gave in the Whatsapp group. Patients who did not respond were called by phone and checked to see if they provided continuity. Both the exercise group and the control group continued their drug treatments during this period.

Group 2: Control group: Individuals in the control group continued their routine drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with rheumatic disease,
* Participants knew the exercises before attending BETY sessions,
* Participants who could participate in telerehabilitation by following WhatsApp communication were included in the exercise group.

Exclusion Criteria:

* Participants with neurological and psychological disorders,
* severe respiratory failure, fractures, infections, cancer, and musculoskeletal pain due to surgery in the last 6 months,
* Vision loss,
* Pregnancy
* Participants who did not agree to volunteer were not included in our study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Health Assessment Questionnaire at 8 weeks | Baseline, 8 weeks
  The Turkish version of the Health Assessment Questionnaire (HAQ), which is frequently used in patients with rheumatism, was used to evaluate their health and disability status.
  This questionnaire consists of 20 questions that collect activities of daily living under 8 activity titles, and each answer is given a score between 0 and 3. (0; No difficulty, 1; With some difficulty, 2: With great difficulty, 3: Not at all).
  To calculate the total score, these scores are added and divided by 8 based on the highest score in all sections. A high score is interpreted negatively.
Change from Baseline in Health Anxiety and Depression Scale at 8 weeks | Baseline, 8 weeks
  The Turkish version of the Health Anxiety and Depression Scale (HADS) was used to evaluate depression and anxiety levels.
  This scale consists of 14 questions, focusing on the last few days. Each question has 4 options. Odd-numbered questions are used for anxiety, even-numbered questions are used to evaluate depression, and 2 separate scores are obtained that can take values between 0-21. While the critical value for anxiety in the sub-title of the scale was 10, it was determined to be 7 for depression.
Change from Baseline in Biopsychosocial Exercise Therapy Questionnaire (BETY-BQ) at 8 weeks | Baseline, 8 weeks
  The Biopsychosocial Exercise Therapy Questionnaire (BETY-BQ), consists of 30 questions. Each of the items in the scale is scored between 0-4 in accordance with the Likert system.
  A higher score indicates poor biopsychosocial status (4: Yes always, 3: Yes often, 2: Yes sometimes, 1: Yes rarely, 0: No, never).

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No